CLINICAL TRIAL: NCT01861353
Title: Randomized Controlled Trial of the Effect of Cranberry-lingonberry Juice on the Occurrence of Urinary Tract Infections, the Gut Microbiota, and the Uropathogenic Escherichia Coli
Brief Title: Cranberry-lingonberry Juice Started During Acute Infection in Prevention of Urinary Tract Infections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, Senior consultant in pediatric infectious diseases, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EETTMK74/2012
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Urinary Tract Infection; Pyelonephritis; Cystitis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis; Cystitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry-lingonberry juice (Experimental): Cranberry-lingonberry juice. Cranberry 12.8%, Lingonberry 12.4%, together 38g/l, contains added sugars 10g/dL.
  Dose is 5 mL/kg/day, max. 300 ml/day per day. Juice was manufactured and donated by Eckes-Granini, Finland
  Interventions: Other: Cranberry-lingonberry juice
- Placebo juice (Placebo Comparator): Contains no cranberry or lingonberry extracts. Added sugars 10g/dL (same as in the active juice group). Contains natural cranberry flavour and red anthocyanin colour. Contains 5.5 g/L citric acid. Has been tested by chemists and does not contains PAC-compounds which are thought to be the main active compound in cranberry juice.
  Placebo juice was manufactured by Eckes-Granini. Dose is 5 mL/kg/day, max. 300 mL/day.
  Interventions: Other: Placebo juice

INTERVENTIONS:
Other: Cranberry-lingonberry juice
  Arms: Cranberry-lingonberry juice
Other: Placebo juice — Juice iwth similar sugar concentration as cranberry-lingonberry juice but without berry extracts
  Arms: Placebo juice

SUMMARY:
Cranberry and cranberry-lingonberry juice prevented urinary tract infections in children and in adults in our earlier clinical trials. The preventive effect was, however, observed late in the follow-up and the next recurrence was not prevented in children. The investigators hypothesize that cranberry-lingonberry juice should be started already during the antimicrobial treatment of acute urinary tract infection in order to maximize the preventive efficacy of the juice. In addition, the investigators aim to find the explanation for the efficacy of cranberry-lingonberry juice by analyzing the concomitant changes in the chemical composition of urine and feces as well as the changes of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Recent confirmed urinary tract infection, diagnosed in Oulu University Hospital or Oulu Health Care Center
* Age 1-16 years

Exclusion Criteria:

* Continuous antimicrobial prophylaxis
* Age < 12 months or > 16 years
* Severe congenital kidney or other urinary tract anomaly in ultrasound

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change of the intestinal and urinary microbiome | 3 months to 12 months

SECONDARY OUTCOMES:
The occurrence of urinary tract infections (infection episodes/person years at risk) | 12 months
Time to the first recurrence | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Jepson RG, Mihaljevic L, Craig JC. Cranberries for treating urinary tract infections. Cochrane Database Syst Rev. 2023 Dec 14;12(12):CD001322. doi: 10.1002/14651858.CD001322.pub2. PMID 38096261
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952